CLINICAL TRIAL: NCT02541747
Title: Assessments in Stress and Quality of Sleep/Life in Night-shift Nurses and Doctors
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Taichung Veterans General Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CG14114
Record Dates: First submitted 2015-06-20; First posted 2015-09-04 (Estimated); Last update posted 2016-07-12 (Estimated); Status verified 2015-09

CONDITIONS: Shift-Work Sleep Disorder
MeSH Terms: conditions — Sleep Disorders, Circadian Rhythm | interventions — Massage

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- massage (Active Comparator): massage for 30 min, once a week for 4 weeks
  Interventions: Behavioral: massage
- control (No Intervention): Rest as control

INTERVENTIONS:
Behavioral: massage — massage
  Arms: massage

SUMMARY:
This study aims to evaluate the effects of aroma massage to sleep quality of the nurses and staff during night shift.

DETAILED DESCRIPTION:
Night shift increases physical and psychological pressure, and even affects their sleep quality. This study aims to evaluate the effects of aroma massage to sleep quality of the nurses during night shift after life-style modification and/or aroma massage. The investigators adopt a Randomized Controlled Trial (RCT) in this study. The investigators expect aroma massage would improve the sleep quality during night shift.

ELIGIBILITY:
Inclusion Criteria:

* Shift-Work Nurses and Staff

Exclusion Criteria:

* Diabetes mellitus, cardiovascular disease and psychological disorders

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 77 (Actual)
Dates: Start 2014-06; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
brain-derived neurotrophic factor | 4 weeks

SECONDARY OUTCOMES:
Pittsburgh sleep quality index (PSQI) | 4 weeks
  Psychological questionnaire
Depression score ( Zung's Self-Reported Depression Scale) | 4 weeks
  Psychological questionnaire- Zung's Self-Reported Depression Scale
Anxiety score (Beck Anxiety Inventory) | 4 weeks
  Psychological questionnaire- Beck Anxiety Inventory
Heart rate variability | 4 weeks
  Cardiopulmonary functions
Metabolic syndrome (NCEP) | 4 weeks
  Third Report of the National Cholesterol Education Program (NCEP) criteria
VCAM-1 | 4 weeks
  Cardiovascular risk and Inflammatory markers
Irisin | 4 weeks
  Cardiovascular risk and Inflammatory markers
circadian rhythm | 4 weeks
  orexin

CONTACTS AND LOCATIONS:
Overall Officials: Wayne HH Sheu, MD, PhD, Principal Investigator — Taichung Veterans General Hospital
Locations (1):
- Division of Endocrinology and Metabolism, Department of Internal Medicine, Taichung Veterans General Hospital, Taichang, Taiwan

IPD SHARING:
Plan to Share IPD: No